CLINICAL TRIAL: NCT07034352
Title: Health Impact 360: Advancing Physical, Social, and Mental Health Among Marginalized Communities for Cardiovascular Health Equity
Acronym: HI360
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Detroit Hispanic Development Corporation (Unknown); Eastside Community Network (Unknown); Community Health and Social Service Center (CHASS) (Unknown)
Responsible Party: Principal Investigator, Jennifer Garner, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00256551; OT2HL158287 (NIH)
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Health Promotion; Cardiovascular Health
Keywords: Health Program; Health outcomes; Black, indigenous, people of color; Social health; Walking; Health Education and support; Mental health; social support
MeSH Terms: conditions — Health Education; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a waitlist-control trial. The intervention-randomized participants will receive the intervention first in "Wave 1" and the participants randomized to the control group, "Wave 2", will experience a delay in access to the program until after the end of the Wave 1 intervention period at each participating site.
Who Masked: Outcomes Assessor
Masking Description: Statisticians will be blinded to arm assignment during analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Impact 360 (Experimental): 16-week, group-based comprehensive health program that covers all behavioral and clinical dimensions of heart health: healthy eating, physical activity, quality sleep, tobacco cessation, blood pressure, cholesterol, Hemoglobin A1c, and Body Mass Index.
  Interventions: Behavioral: Health Impact 360
- Usual care - Wait list control (Other): Participants that will be on the wait list will be evaluated. These participants will be enrolled into the treatment program 16-20 weeks after the first treatment group.
  Interventions: Other: Usual care - Wait list control

INTERVENTIONS:
Behavioral: Health Impact 360 — Participants will be assigned to a team and teams will meet 1-2 times per week for sessions at a local community organization. Sessions will be up to 2 hours long and will include two parts: (1) 30-60 minutes of activities related to physical, mental, social, financial, and community health, and (2) 60-75 minutes of group physical activity (walking), including stretches to warm up and cool down.
  Arms: Health Impact 360
Other: Usual care - Wait list control — Participants will be on this for approximately 16 weeks and be asked to complete data collection information at baseline and 16 weeks.
  Arms: Usual care - Wait list control

SUMMARY:
The purpose of this clinical trial is to evaluate an evidence-based intervention, Health Impact 360, toward the promotion of cardiovascular health (CVH), including physical, mental, and social health outcomes, among adults living in marginalized communities.

Study hypotheses include:

* Participants in the Health Impact 360 intervention arm will have better CVH (i.e., a higher overall LE8 score) at the 16-week endpoint compared to the control.
* Participants in the Health Impact 360 intervention arm will report better mental health (i.e., a lower perceived stress score) at the 16-week endpoint compared to the control.
* Participants in the Health Impact 360 intervention arm will report better social support and well-being (i.e., higher emotional support and instrumental support scores and reduced social isolation) at the 16-week endpoint compared to control.
* Participants with greater intervention engagement (e.g., better session attendance) will experience greater intervention impacts across all primary and secondary outcomes relative to the minimally engaged peers.

Researchers will compare outcomes among intervention participants to outcomes among delayed intervention control participants who will be invited to participate in Health Impact 360 once all endpoint measures are collected.

Participants will:

* Engage in group-based programming twice per week for 8 weeks
* Engage in group-based programming once per week for 8 weeks
* Participate in survey-based and biometric data collection at two timepoints: baseline and 16-week endpoint
* Self-monitor their physical activity via a study-provided pedometer

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Able to participate in group-based programming

Exclusion Criteria:

- All pregnant persons to prevent pregnancy-related biometric changes from biasing outcome analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiovascular health (CVH) based on the Life's Essential 8 score (LE8) | Baseline, 16 weeks
  LE8 CVH Score will be averaged for each participant at baseline and 16 weeks on the individual LE8 metrics (i.e., scores of 0-100 for eight items). An average score of 0 to 49 is defined as low CVH, 50 to 79 is moderate CVH, and 80 to 100 is high CVH.

SECONDARY OUTCOMES:
Change in mental health based on the perceived stress scale | Baseline, 16 weeks
  The Perceived Stress Scale (PSS) is a 10-item scale that was developed to measure the degree to which situations in one's life are appraised as stressful. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Scores range from 0 to 40 with higher scores indicating a worse outcome.
Change in social health via the 4-item Patient-Reported Outcomes Measurement Information System (PROMIS) emotional support scale | Baseline, 16 weeks
  This is a 4-item survey that participants select from never (1) - always (5). The score range is from 4-20 with a higher score indicating more emotional support.
Change in social health via the 4-item Patient-Reported Outcomes Measurement Information System (PROMIS) instrumental support scale | Baseline, 16 weeks
  This is a 4-item survey that participants select from never (1) - always (5). The score range is from 4-20 with a higher score indicating more instrumental support.
Change in social health via the 4-item Patient-Reported Outcomes Measurement Information System (PROMIS) social isolation scale | Baseline, 16 weeks
  This is a 4-item survey that participants select from never (1) - always (5). The score range is from 4-20 with a higher score indicating greater social isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Garner, PhD, RD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Community Health and Social Service Centers (CHASS), Detroit, Michigan
  - Eastside Community Network (ECN), Detroit, Michigan
  - Detroit Hispanic Development Corporation (DHDC), Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available as soon as the primary team has completed the analysis as proposed in the grant, and no later than time of an associated publication or end of the grant award, whichever comes first. Data deposited in Deep Blue Data will be accessible for at least 10 years, after which it will be appraised for continued preservation by University Library personnel.
Supporting Information: Study Protocol, ICF
Time Frame: Data deposited in Deep Blue Data will be accessible for at least 10 years, after which it will be appraised for continued preservation by University Library personnel.